CLINICAL TRIAL: NCT04362215
Title: Heart Aging When Near Vision Difficulty Begins
Status: Completed | Type: Observational
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Şahbender Koç, Principal Investigator, Kecioren Education and Training Hospital
Other Study IDs: 09/2019/1953
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Aging
Keywords: aging; heart aging; presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- High AA group: Group 1 consisted of those having an AA level of 3.57-4.16 D (high AA group; those who had near clear vision between 24-28 cm). .
  Interventions: Diagnostic Test: Subjective accomodation amplitude measurement
- Low AA group: Group 2 consisted of those having an AA level of 3.44-3.03 D (low AA group; those who had near clear vision between 29-33 cm)
  Interventions: Diagnostic Test: Subjective accomodation amplitude measurement

INTERVENTIONS:
Diagnostic Test: Subjective accomodation amplitude measurement — ECG:Electrocardıography Echocardiography, Holter implementation(for Lf/Hf ratio))
  Other Names: ECG,Echocardiography,Holter implementation

SUMMARY:
Near vision deterioration during aging results from a decrease in accomodation amplitude (AA). Myocardial regeneration is limited, and cardiac aging is an independent risk factor for cardiovascular disease. Thus, the investigators investigated the association between cardiac aging and AA.

The subjects (500, mean 50-year-old subjects, with equal males and females) were divided into two groups according to AA measured with a Raf ruler. Biomicroscopy was used to capture images of the lens nucleus in the unaccommodated state, followed by images of a 4 diopter (D) accommodated state. The nucleus diameter change at 1 D accomodation was measured using ImageJ. Cardiac conduction system differences were evaluated using electrocardiography, and cardiac autonomic aging was assessed based on heart rate variability. Myocardial aging was assessed based on diastolic dysfunction.

DETAILED DESCRIPTION:
Lens cells and proteins are encapsulated, and they are not turned over or replaced.The lens nucleus starts to form before birth, so the nucleus is one of the three oldest tissues in the body .With aging, continuous cardiomyocyte stress derails proteostasis by causing excessive autophagy and protease activation, and, ultimately, contractile and electrophysiological dysfunction. Aggregate deposition, proteostasis deterioration, and diffusion degradation between the nucleus and cortex are the main reasons for lens aging.Heart, lens, and neuronal cells change significantly with age, and they are older than cells from renewable tissues.

Near vision deterioration during aging results from a decrease in accomodation amplitude (AA). Cardiac aging is an independent risk factor for cardiovascular disease. Thus, the investigators investigated the association between cardiac aging and AA. The subjects (500 mean 50-year-old subjects, with equal males and females) were divided into two groups according to AA measured with a Raf ruler. The nucleus diameter change at 1 D accomodation was measured using ImageJ. Cardiac conduction system differences, autonomic aging, myocardial aging were evaluated using electrocardiography, heart rate variability and diastolic dysfunction. For near distance vision,compared to subjects who could see clearly from 24-28 cm, subjects who could see clearly from 29-33 cm had a 2.104-fold higher risk of a lateral e' velocity <10 cm/s[95%CI; 1.312-3.374], 2.603-fold higher risk of diastolic dysfunction[95%CI; 1.453-4.662], 1.54-fold higher risk of a low/high frequency ratio >3.1, [95%CI;1.085-2.197]. Subjective AA measurement can predict important heart aging parameters.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers, mean 50 years of age (49-51)

Exclusion Criteria:

Hypertension, Diabetes mellitus, Atrial fibrillation, Coronary artery disease, Arrhythmia, Hyperthyroidism , Anemia, Heart failure, Respiratory diseases, Severe obesity (body mass index ≥35 kg/m2),

Ages: 49 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers ,mean 50 years of age (49-51)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
ECG interval changes meauserements(ms,mm,number) | 1 day
  ECG PR interval (ms),Ventricle Premature Systol(number),Left Ventricle Hypertrophy(mm)Right Bundle Branch,Left Bundle Branch (the presence / absence)
Holter implementation | 1 day
  To detect autonomic cardiac aging based on heart rate variability (HRV),the low frequency (LF)/high frequency (HF) ratio was measured using a CardioScan II (version 11.4.0054a; DMS Software, Stateline, NV, USA)
Echocardiographic measurements | 1 day
  Diastolic dysfunction meauserements(mitral anulus lateral e' velocity <10 cm/s, average E/e' ratio >14, Left atrium maximum volume index (LAv.i.) >34 mL/m2, and peak Tricuspit Regurgitation velocity >2.8 m/s.

CONTACTS AND LOCATIONS:
Overall Officials: Şahbender Koç, Principal Investigator — University of Health Sciences Ankara Keçiören Education Hospital
Locations (1):
- ANkara Keçiören EAH, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Koc S, Baysal SS. Heart aging when near vision difficulty begins. Aging Male. 2020 Dec;23(5):1346-1354. doi: 10.1080/13685538.2020.1766438. Epub 2020 May 25. PMID 32449445